CLINICAL TRIAL: NCT03469375
Title: Modified-FOLFIRINOX Regimen Based Neoadjuvant Therapy in Chinese Patients With Locally Advanced Pancreatic Cancer
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: SAHZhejiangU-FOL
Record Dates: First submitted 2018-03-12; First posted 2018-03-19 (Actual); Last update posted 2018-03-27 (Actual); Status verified 2014-04

CONDITIONS: Pancreatic Cancer; Chemotherapy Effect; Surgery--Complications
Keywords: FOLFIRINOX; Pancreatic cancer; Conversion surgery; Overall survival
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Neoadjuvant Therapy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- LAPC patients with mFOFLRINOX-based neoadjuvant therapy: LAPC patients were enrolled prospectively and diagnosed by MDT group in our hospital. These patients further received the neoadjuvant therapy with mFOLFIRINOX, the Overall survival, Progression survival, response to mFOLFIRINOX, chemo-related Toxicities, Postoperative complications and Histopathologic staging were measured.
  Interventions: Drug: modified-FOLFIRINOX

INTERVENTIONS:
Drug: modified-FOLFIRINOX — LAPC patients with mFOLFIRINOX-based neoadjuvant therapy or not was set as the main intervention
  Other Names: Neoadjuvant therapy

SUMMARY:
FOLFIRINOX regimen is first-line neoadjuvant chemotherapies for patients with locally advanced pancreatic cancer (LAPC) worldwide. However, FOLFIRINOX is not well accepted in China because of the high prevalence of adverse events and poor tolerance. To evaluate the safety and efficacy of modified-FOLFIRINOX (mFOLFIRINOX) in Chinese LAPC patients and compare survival between LAPC patients with mFOLFIRINOX-based preoperative therapy and LAPC patients who underwent surgery alone.

DETAILED DESCRIPTION:
At this institution, a mFOLFIRINOX regimen has been adopted for metastatic pancreatic cancer (MPC) patients and promising results obtained. The modification resulted in a significantly reduced prevalence of severe adverse events in MPC patients, whereas the OS and PFS were extended to 10.3m and 7.0m, respectively, which is similar to that for patients on a full-dose regimen. Therefore, the investigators further evaluated the efficacy of mFOLFIRINOX in LAPC patients. Here, investigators want to prospectively enroll LAPC patients who underwent preoperative therapy with mFOLFIRINOX from April 2014 and compared the surgical resectability and surgical morbidity/surgical mortality among patients with surgically resectable pancreatic cancer (RPC) or LAPC who underwent surgery alone retrospectively. For patients with LAPC, mFOLFIRINOX was administrated for several cycles until the optimal response was obtained and then patients were evaluated for surgery. Moreover, survival data, including OS and PFS, were determined.

ELIGIBILITY:
Inclusion Criteria:

1. The patients are diagnosed by histology to have pancreatic adenocarcinoma
2. The patients are defined as locally advanced pancreatic cancer according to NCCN guideline
3. The patients prescribed mFOLFIRINOX-based neoadjuvant therapy

Exclusion Criteria:

1. ECOG performance score more than 2
2. Insufficient bone marrow, liver and renal function
3. Patients with other malignancies
4. Patients were older than 85 years or less than 18 years

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All locally advanced pancreatic cancer (LAPC) patients are diagnosed by histology to have pancreatic adenocarcinoma after a biopsy and prescribed mFOLFIRINOX-based neoadjuvant therapy at the Department of Hepatobiliary and Pancreatic Surgery of the Second Affiliated Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2014-04-01 (Actual); Primary Completion 2017-11-01 (Actual); Study Completion 2017-11-01 (Actual)

PRIMARY OUTCOMES:
Overall survival | 2014-04-01 to 2017-11-01
  the duration from the date of hospital admission to death of any cause.
Progression free survival | 2014-04-01 to 2017-11-01
  the duration from the date of hospital admission to disease progression or death.

SECONDARY OUTCOMES:
Response to mFOLFIRINOX | 2014-04-01 to 2017-11-01
mFOLFIRINOX related adverse events | 2014-04-01 to 2017-11-01
Postoperative complications | 2014-04-01 to 2017-11-01
Histopathologic staging | 2014-04-01 to 2017-11-01

CONTACTS AND LOCATIONS:
Locations (1):
- the second affiliated hospital of Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided